CLINICAL TRIAL: NCT02465164
Title: Cervical Ripening With Cook Catheter Plus Low Dose Oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Justin Bruner, Resident Physician, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HFM 2900
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Cervical Ripening
MeSH Terms: interventions — Oxytocin

ARMS (2):
- Cook catheter (Other): Control
  Interventions: Device: Cook catheter
- Cook catheter plus low dose oxytocin (Active Comparator): Test group
  Interventions: Device: Cook catheter; Drug: Oxytocin

INTERVENTIONS:
Device: Cook catheter
Drug: Oxytocin
  Arms: Cook catheter plus low dose oxytocin

SUMMARY:
The purpose of this study is to compare if using a Cook Cervical Ripening Balloon in conjunction with low dose oxytocin is more effective at shortening labor induction times than the Cook Cervical Ripening Balloon alone. After obtaining consent, patients will be randomly divided into a Balloon with oxytocin or Balloon only group. The Balloon will be placed by either Resident or Attending Physicians and left in place for 12 hours (protocol) in both groups or until it falls out. After either 12 hours or the Balloon falls out, oxytocin will be used for the remainder of the induction per current hospital protocol. Time to delivery, mode of delivery, average number of hours Balloon remained in place, non-reassuring fetal heart tracings, adverse outcomes (ie fetal malpresentation, postpartum hemorrhage) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy
2. reassuring fetal status at time of presentation
3. Bishop Score <6

Exclusion Criteria:

1. Closed cervix
2. Breech presentation
3. Multiple gestations
4. Recent vaginal bleeding
5. Placenta previa
6. non reassuring fetal status
7. Active genital herpes infection

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Cook Catheter: Control
  Cook catheter
- Cook Catheter Plus Low Dose Oxytocin: Test group
  Cook catheter
  Oxytocin
Period: Overall Study
Arm/Group | Cook Catheter | Cook Catheter Plus Low Dose Oxytocin
Started | 16 | 10
Completed | 16 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cook Catheter | Cook Catheter Plus Low Dose Oxytocin | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (1.2) | 24 (1.3) | 23 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery (in Hours)
Description: Cook Only group Cook + Pitocin group N Mean (hrs) (SD) 16 27.9 (9.6) 10 23 14.6)
Time Frame: Up to 60 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Cook Catheter | Cook Catheter Plus Low Dose Oxytocin
Number analyzed (Participants) | 16 | 10
hours | 27 [12 to 54] | 23 [7 to 33]
Statistical Analysis 1: Comparison: Cook Catheter vs Cook Catheter Plus Low Dose Oxytocin; Test type: Other — Wilcoxon rank-sum tests; p = 0.208, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Cook Catheter | Cook Catheter Plus Low Dose Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes